CLINICAL TRIAL: NCT02193984
Title: Alliance to Control Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: San Diego State University (Other)
Collaborators: Peers for Progress (Other); American Academy of Family Physicians (Other)
Responsible Party: Principal Investigator, Guadalupe X. Ayala, Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: G00007943
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; Peer support; Hispanic; Latino
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peer support (Experimental): Study participants are assigned a volunteer peer supporter who has been trained to offer support on diabetes management.
  Interventions: Behavioral: Peer support
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Peer support
  Arms: Peer support

SUMMARY:
Alliance to Control Diabetes was a 2.5-year study funded by the American Academy of Family Physicians Foundation. The study was designed to help patients better manage their diabetes, and was a partnership between the Institute for Behavioral and Community Health and Clínicas de Salud del Pueblo, Inc (CDSDP), a private, non-profit corporation providing comprehensive primary care services to residents throughout Imperial and Riverside Counties, California. The investigators identified 336 patients with uncontrolled diabetes from three CDSDP clinics. Patients were randomly assigned to intervention or control conditions. The 12-month intervention consisted of individual diabetes management support delivered by a trained volunteer peer supporter. The primary aim was determine if peer support can help patients better manage their diabetes and improve the quality of their lives. Intervention effectiveness was evaluated through volunteer and patient surveys at baseline, 6 months and 12 months. This study was part of the global Peers for Progress network which has been testing peer support programs in 13 countries.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years old
* Must be diagnosed with Diabetes Mellitus Type I, Diabetes Mellitus Type II or Gestational Diabetes
* Must be a resident of Imperial County
* Must be a current patient of Clínicas de Salud del Pueblo, Inc., at one of the three participating clinics
* Must speak Spanish and/or English
* Must plan on remaining in Imperial County for at least 12 months after enrollment into the study

Exclusion Criteria:

* Must not be involved in any other diabetes-related study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2009-02; Primary Completion 2012-01 (Actual); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Changes in HbA1c levels. | Baseline, 6 months, 12 months
  Changes in HbA1c levels of diabetes patients from baseline to 12 months as assessed by medical chart review of blood draw results.

SECONDARY OUTCOMES:
Changes in blood pressure. | Baseline, 6 months, 12 months
  Changes in blood pressure of diabetes patients from baseline to 12 months as assessed by medical chart review.
Changes in cholesterol. | Baseline, 6 months, 12 months
  Changes in cholesterol of diabetes patients from baseline to 12 months as assessed by medical chart review.
Changes in HDL, LDL and triglycerides. | Baseline, 6 months, 12 months
  Changes in HDL, LDL and triglycerides of diabetes patients from baseline to 12 months as assessed by medical chart review.
Changes in depression. | Baseline, 6 months, 12 months
  Changes in depression of diabetes patients from baseline to 12 months as assessed by self-report via interview with a trained research assistant in the participant's language of choice (Spanish or English).
Changes in distress. | Baseline, 6 months, 12 months
  Changes in distress of diabetes patients from baseline to 12 months as assessed by self-report via interview with a trained research assistant in the participant's language of choice (Spanish or English).

CONTACTS AND LOCATIONS:
Overall Officials: Guadalupe X Ayala, PhD, MPH, Principal Investigator — San Diego State University
Locations (2):
- United States (2):
  - San Diego State University Research Foundation, Calexico, California
  - San Diego State University Research Foundation, San Diego, California

REFERENCES:
- [Background] Fisher EB, Ayala GX, Ibarra L, Cherrington AL, Elder JP, Tang TS, Heisler M, Safford MM, Simmons D; Peers for Progress Investigator Group. Contributions of Peer Support to Health, Health Care, and Prevention: Papers from Peers for Progress. Ann Fam Med. 2015 Aug;13 Suppl 1(Suppl 1):S2-8. doi: 10.1370/afm.1852. PMID 26304968
- [Background] Simmons D, Bunn C, Nakwagala F, Safford MM, Ayala GX, Riddell M, Graffy J, Fisher EB. Challenges in the Ethical Review of Peer Support Interventions. Ann Fam Med. 2015 Aug;13 Suppl 1(Suppl 1):S79-86. doi: 10.1370/afm.1803. PMID 26304976
- [Result] Parada H Jr, Horton LA, Cherrington A, Ibarra L, Ayala GX. Correlates of medication nonadherence among Latinos with type 2 diabetes. Diabetes Educ. 2012 Jul-Aug;38(4):552-61. doi: 10.1177/0145721712445215. Epub 2012 Apr 30. PMID 22546741
- [Result] Ayala GX, Ibarra L, Cherrington AL, Parada H, Horton L, Ji M, Elder JP. Puentes hacia una mejor vida (Bridges to a Better Life): Outcome of a Diabetes Control Peer Support Intervention. Ann Fam Med. 2015 Aug;13 Suppl 1(Suppl 1):S9-17. doi: 10.1370/afm.1807. PMID 26304977
- [Result] Soto SC, Louie SY, Cherrington AL, Parada H, Horton LA, Ayala GX. An ecological perspective on diabetes self-care support, self-management behaviors, and hemoglobin A1C among Latinos. Diabetes Educ. 2015 Apr;41(2):214-23. doi: 10.1177/0145721715569078. Epub 2015 Feb 5. PMID 25656696
- See also: Related Info — http://www.peersforprogress.org